CLINICAL TRIAL: NCT06172530
Title: Observational Study on the Improvement of Dry Eye Syndrome, Treatment Satisfaction, and Intraocular Tolerance With Diquasol Eye Drops and Hyaluron/Hyaluronmax Eye Drops in Patients Over 19 Years Old With Dry Eye Syndrome
Brief Title: Observational Study on the Improvement of Dry Eye Syndrome, Treatment Satisfaction, and Intraocular Tolerance With Diquasol Eye Drops
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: HL-DQAS-401
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-11

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is to verify the efficacy and safety in the treatment of dry eye syndrome in patients prescribed with Diquasol eye drops as a monotherapy, or in combination with Hyaluron eye drops, or in combination with Hyaluronmax eye drops.

DETAILED DESCRIPTION:
This study is to observe the prescription patterns in routine clinical practice and assess the changes in dry eye symptoms, treatment satisfaction, and intraocular tolerance over a 12-week period in patients prescribed with Diquasol eye drops as a monotherapy or in combination with Hyaluron eye drops or Hyaluronmax eye drops for the treatment of dry eye syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years and older
* Patients with dry eye syndrome with TBUT of 10 or less
* Individuals scheduled to receive either Diquasol eye drops as a monotherapy or a combination therapy of Diquasol eye drops with Hyaluron eye drops or Diquasol eye drops with Hyaluronmax eye drops, based on clinical judgment for the treatment of dry eye syndrome
* Individuals who have voluntarily provided written consent for participation in this study

Exclusion Criteria:

* Pregnant or lactating women
* Individuals contraindicated according to the approval conditions of Diquasol eye drops, Hyaluron eye drops, and Hyaluronmax eye drops
* Cases where the principal investigator or study personnel deem the individual unsuitable for participation in this clinical study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dry eye syndrom patients aged 19 years or older
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Primary Assessment Variables | after 12 weeks of prescription for Diquasol eye drops and Hyaluron/Hyaluronmax eye drops compared to baseline
  Changes in Tear Break-Up Time (TBUT) after 12 weeks according to each group, including monotherapy with Diquasol eye drops, combination therapy with Diquasol eye drops and Hyaluron eye drops, and combination therapy with Diquasol eye drops and Hyaluronmax eye drops.

CONTACTS AND LOCATIONS:
Overall Officials: ChounKi Joo, Principal Investigator — CK st. Mary's Eye Clinic
Locations (1):
- CK St. Mary's Eye Clinic, Seoul, South Korea